CLINICAL TRIAL: NCT01777958
Title: Noninterventional Study - Advanced HER2-positive Breast Cancer (Metastatic or Locally Recurrent, Inoperable): First-Line Treatment With PERJETA After Adjuvant Herceptin Therapy (HELENA)
Brief Title: HELENA Study: An Observational Study of Perjeta (Pertuzumab) in First-Line Treatment in Patients With Her2-Positive Advanced Breast Cancer After Adjuvant Herceptin Therapy
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28750
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the efficacy, safety and patient reported quality of life of palliative first-line Perjeta (pertuzumab) in combination with Herceptin (trastuzumab) in patients with HER2-positive advanced breast cancer (metastatic or locally recurrent, inoperable) who relapsed after completed adjuvant Herceptin therapy. Additionally, information on selection criteria of breast cancer patients treated first-line with Perjeta, Herceptin and chemotherapy and their treatment duration will be collected and analyzed. Data will be collected from eligible patients for up to 20 months of treatment and 24 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female adult patients, >/= 18 years of age
* HER2-positive advanced breast cancer (metastatic or locally recurrent, inoperable) relapsing after completed adjuvant Herceptin therapy
* Indication for first-line treatment with Perjeta in combination with Herceptin and chemotherapy according to the Summary of Product Characteristics
* Prior Herceptin therapy as systemic adjuvant treatment (postoperative treatment in a potentially curable setting); additional upfront neoadjuvant Herceptin therapy is allowed
* No prior chemotherapy and/or immunotherapy for advanced (metastatic or locally recurrent, inoperable) HER2-positive breast cancer

Exclusion Criteria:

* Pregnant or breastfeeding women
* Contraindications to Perjeta, Herceptin or concomitant chemotherapy according to the Summary of Product Characteristics
* No Herceptin treatment for early breast cancer in the adjuvant setting

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with HER2-positive advanced breast cancer (metastatic or locally recurrent, inoperable)who relapsed after adjuvant Herceptin therapy, with indication for treatment with Perjeta in combination with Herceptin
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2013-06-14 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Median progression-free survival in routine clinical practice | approximately 7.5 years

SECONDARY OUTCOMES:
Dosage/schedule: Initiation/duration/modification/discontinuation of Perjeta administration | approximately 7.5 years
Clinical/demographic patients characteristics at initiation of treatment | approximately 7.5 years
Safety: Incidence of adverse events | approximately 7.5 years
Patient reported outcome: Quality of life (FACT B questionnaire) | approximately 7.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- AGAPLESION Markus-Krankenhaus, Frankfurt, Germany